CLINICAL TRIAL: NCT04890899
Title: Splenic Preserving Surgery in Hydatid Spleen
Brief Title: Splenic Surgery for Hydatid Spleen in Single Institutional Experience
Status: Completed | Type: Observational
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JabirIbnHayyanMU
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Spleen; Cyst, Hydatid (Manifestation)
Keywords: Spleen; Hydatid cyst; Surgery; Preserving surgery
MeSH Terms: conditions — Cysts; Echinococcosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cystic enculation of spleen hydatid — Preoperative preparation did according to the general condition of the patient and fitness for anaesthesia. Laparotomy did under general anaesthesia, supine position, the abdomen opened either by midline or left subcostal incision. Identification of splenic hydatid cyst. Exploration of the peritoneal cavity for undetected hepatic or peritoneal hydatid preoperatively. Isolation of operative field by packs socked with hypertonic solution (20 -30 % hypertonic saline). Aspiration of the cyst fluid. Injection of suitable amount about 5 ml of (1 % of cetramid) solution and waiting for at least 5 minutes and then re-aspiration. The spleen is not needed to mobilize. Extraction of the endocyst and washing of the cavity with normal saline. Occupying the cystic cavity intracystic drain. Perioperative and postoperative close observation of the patient for an anaphylactic reaction or any other complication. Follow-up of the patient until discharge from hospital on (3th - 5th) days.

SUMMARY:
Splenic-preserving surgery in hydatid spleen: Single intuitional experience

DETAILED DESCRIPTION:
Background:

Although hydatid disease affects many organs in the human body, splenic hydatid represents about 0.8-4% of all human echinococcosis cases. Until recently, splenectomy was the recommended surgical procedure for splenic hydatid. Since 1980 there has been an increasing tendency to use conservative option to deal with such pathology.

Aim of the study:

To evaluate our experience in open splenic-preserving surgery for splenic hydatid in a single institutional study.

Patient and methods:

A retrospective study. Ten patients with splenic hydatid were operated upon from August 2013 to January 2018 in our medical centre. Spleen has affected alone in 7 cases, liver and spleen were affected in 3 cases, and one of them had intraperitoneal cyst affection in addition. The diagnosis confirmed mainly by ultrasonography. In some cases, it computed tomography CT scan, and magnetic resonance imaging MRI were needed. Chest X-ray had taken for all patients to exclude pulmonary hydatid. The open surgical procedure used. Isolation of the field, aspiration of cystic fluid and injection of 1% cetrimide solution, re-aspiration, endocystectomy, suturing of cystic edges over intracystic tube drain. All surgery did under cover of albendazole pre and postoperative 15mg/kg/day.

Results:

No significant intraoperative and postoperative complications. No reoperation was needed. Hospital stays 3-5 days. No recurrence after (1-3) year follow-up. However, three patients missed follow-up after two years.

Conclusion:

Our experience in splenic hydatid encourages us to use splenic-preserving surgery whenever possible instead of splenectomy.

ELIGIBILITY:
Inclusion Criteria:

Single hydatid spleen Primary spleen hydatid

-

Exclusion Criteria:

* Multiple splenic hydatid Rupture hydatid spleen

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: from 5- 40 years (mean 23.6 years).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
splenic sparing surgery for hydatid spleen | 3 year
  Six of them males and four females, their age range from 5- 40 years (mean 23.6 years). Hydatid spleen alone was found in seven cases while splenic and liver hydatid was found in three cases one of them had peritoneal hydatid affection in addition. Hospital stay was ranged from 3-5 days.

IPD SHARING:
Plan to Share IPD: Yes
Splenic surgery for hydatid spleen, preserve the spleen
Time Frame: 3 years
Access Criteria: documents